CLINICAL TRIAL: NCT00863005
Title: Assessment of the Effects on Barrier Impairment, Clinical Features and Bacterial Colonization of Topical Formulations in Patients With Atopic Eczema; a Phase IIa, Single-center, Randomized, Observer-blind Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Model: Parallel
Other Study IDs: K201-I/280301BS
Record Dates: First submitted 2009-03-12; First posted 2009-03-17 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — K201 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. K201 (Experimental)
  Interventions: Drug: K201
- 2. (Active Comparator)
  Interventions: Drug: K201

INTERVENTIONS:
Drug: K201 — Cream
Drug: K201

SUMMARY:
The purpose of the study is the assessment of the barrier impairment, clinical skin condition and bacterial colonization status in patients with atopic eczema following topical treatment with K201 cream and a comparator twice daily over a 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent obtained;
* male or female patients, 18 years or older;
* manifest atopic eczema diagnosed according to Hanifin and Rajka;
* two comparable lesional areas of 20 - 50 cm2 with a distance of at least 5 cm, clinical condition of atopic eczema mild to moderate (meeting Hanifin and Rajka´s criteria;
* TEWL in the lesional areas at least 12 g/m²h, TEWL value differences ≤ 30 % are allowed between both lesional areas;
* the physical examination must be without disease findings unless the investigator considers an abnormality to be irrelevant to the outcome of the study;
* sexually active females of childbearing potential should either be surgically sterile hysterectomy or tubal ligation), or should use a medically accepted contraceptive regimen:systemic contraceptive (oral, implant, injection), diaphragm or cervical cap with intravaginal spermicide, intrauterine device (IUD), condom with intravaginal spermicide.

Exclusion Criteria:

* acne, eczema other than atopic eczema, hyper- or hypopigmentation or tattoos in the treatment areas;
* suntan which in the opinion of the investigator prevents correct assessments
* dark-skinned persons whose skin color prevents ready assessment of skin reactions;
* evidence of drug or alcohol abuse;
* pregnancy or nursing;
* UV-therapy within 6 weeks before first treatment;
* participation in another clinical study involving pharmaceutical products in the 28 days preceding or during the study;
* symptoms of a clinically significant illness that may influence the outcome of the study in the four weeks before and during the study;
* known allergic reactions to components of the study preparation and the comparator;
* treatment with systemic or locally acting medications which might counter or influence the study aim (e.g. antihistamines or glucocorticosteroids) within two weeks before the beginning of the study (exception: asthma may be found in patients with atopic eczema,therefore inhalation with corticosteroids in patients with asthma accompanying atopic eczema will be allowed at a dose not exceeding 1 mg/day. The dosage should remain constant throughout the study period);
* in the opinion of the investigator or physician performing the initial examination the patient should not participate in the study, e.g. due to probable noncompliance or inability to understand the study and give adequately informed consent;
* patient is institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Transepidermal water loss (TEWL), clinical assessments, corneometry, bacterial counts | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- bioskin GmbH, Hamburg, Germany